CLINICAL TRIAL: NCT05404152
Title: Evaluation of Cognitive Impairment in the Elderly Admitted to Nursing Homes
Status: Completed | Type: Observational
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, MARIA ELENA MOSQUERA LOSADA, Principal Investigator, Universidad de Murcia
Other Study IDs: CIE/UM22
Record Dates: First submitted 2022-05-30; First posted 2022-06-03 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-05

CONDITIONS: Neurocognitive Disorder, Etiology of Neurocognitive Disorder
Keywords: Cognitive impairment, nursing home, neurocognitive disorder
MeSH Terms: conditions — Neurocognitive Disorders; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ederly: Elderly Admitted to Nursing homes

SUMMARY:
This research aims at analysing the profile of the elderly with cognitive impairment (IC) and inquiring about the mental illnesses that cause cognitive impairment of a population (elderly admitted to nursing homes with a high incidence).

DETAILED DESCRIPTION:
The objectives of these studies are to determine the presence of IC and the profile of users who suffer from it in 8 nursing homes in the province of Pontevedra of new admission in 2017, as well as the identification of the frequency of underdiagnosis in the filiation of the mental pathology that causes IC and if that underdiagnosis is related to the presence of doctors or nurses specialists in geriatrics. Sociodemographic, clinical (with special relevance in cognitive assessment and the presence of mental disorders) and functional variables will be analyzed. In addition to providing information that can improve the DC early detection as well as the scarcity of studies in this field, the importance of this research is justified by developing treatment guidelines for people with IC in the future

ELIGIBILITY:
Inclusion Criteria:

* Vounteer
* Elderly Admitted to Nursing homes
* From 60 years old

Exclusion Criteria:

* Elderly without cognitive assessment at admission
* Existence of doubts about the presence of IC

Min Age: 60 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: * Elderly without cognitive assessment at admission
  * Existence of doubts about the presence of IC
Sampling Method: Non-Probability Sample
Enrollment: 390 (Actual)
Dates: Start 2021-12-31 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Study of Evaluation of Cognitive Impairment. MEC o MMSE <24 points or diagnosis of Neurocognitive disorder | Two years

SECONDARY OUTCOMES:
Statistical correlation of CI with educational level. | Two years

OTHER OUTCOMES:
Causes underdiagnosis of IC affiliation and Mental illnesses that cause IC | Two years

CONTACTS AND LOCATIONS:
Overall Officials: MARIA ELENA MOSQUERA LOSADA, MSc in Nursing, Principal Investigator — Universidad de Murcia; ANTONIA GOMEZ-CONESA, PhD, PT, Study Director — Universidad de Murcia; RAMON GONZALEZ CABANACH, PhD, Study Director — Universidade da Coruña
Locations (1):
- UMurcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: Yes